CLINICAL TRIAL: NCT02052596
Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A When Co-administered With Boostrix® in Adults Aged 50 Years and Older
Brief Title: Study to Assess the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine (GSK1437173A) When Co-administered With GSK Biologicals' Diphtheria, Tetanus and Pertussis Vaccine (Boostrix®) in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116887
Record Dates: First submitted 2014-01-23; First posted 2014-02-03 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2017-09

CONDITIONS: Herpes Zoster
Keywords: Boostrix; Herpes zoster; Immunogenicity; Co-administration; Adults; Safety
MeSH Terms: conditions — Herpes Zoster | interventions — Boostrix

ARMS (2):
- GSK1437173A Group (Experimental): Subjects received one injection of Boostrix vaccine and one injection of the GSK1437173A vaccine during the first visit and a second injection of the GSK1437173A vaccine during the third visit, two months later.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: Boostrix
- Control Group (Active Comparator): Subjects received all vaccines separately i.e. one injection of Boostrix vaccine at the first visit, one injection of the GSK1437173A vaccine at the third visit and a second injection of the GSK1437173A vaccine at the fourth visit, all two months apart.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: Boostrix

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK 1437173A — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm at Visit Day 0 and Visit Month 2 for Co-Ad group and at Visit Month 2 and Visit Month 4 for Control group.
Biological: Boostrix — 1 dose administered intramuscularly (IM) in the deltoid region of the dominant arm at Visit Day 0 for both Co-Ad and Control groups.

SUMMARY:
The purpose of this study is to assess immunogenicity, reactogenicity and safety of GSK Biologicals' HZ/su vaccine when its first dose is co-administered with the Boostrix® vaccine in adults aged 50 years or older compared to administration of vaccines separately.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female aged 50 years or older at the time of the first vaccination with the study vaccine(s).
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent). A prednisone dose of < 20 mg/day is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose of study vaccine(s) and ending 30 days after the last dose of study vaccine. This includes any type of vaccine such as (but not limited to) live, inactivated and subunit vaccines (e.g., inactivated and subunit influenza vaccines).
* Administration of long-acting immune-modifying drugs (e.g. infliximab) within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against VZV or HZ and/or planned administration during the study of an HZ or VZV vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* History of HZ.
* Vaccination against diphtheria, or tetanus in the last five years or planned vaccination against diphtheria or tetanus during the study period, other than the study vaccine(s).
* Administration of a combined tetanus, diphtheria and pertussis (Tdap) vaccine at any time prior to study entry.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines including prior severe allergic reaction following tetanus-toxoid, diphtheria-toxoid or pertussis-containing vaccine.
* Hypersensitivity to latex. Note: The investigational HZ/su vaccine does not contain latex.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F by oral route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before 2 months after the last dose of study vaccine.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Any condition which, in the judgment of the investigator, would make intramuscular (IM) injection unsafe.
* Encephalopathy (e.g. coma, decreased consciousness, prolonged seizures) not attributable to an identifiable cause within 7 days of administration of a previous pertussis antigen-containing vaccine.
* Progressive or unstable neurologic disorder.
* History of Arthus-type hypersensitivity reaction following a prior dose of a tetanus-toxoid containing vaccine within the last 10 years.
* History of Guillain-Barré syndrome within 6 weeks of receipt of a prior vaccine containing tetanus toxoid.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 935 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2016-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Lewiston, Maine
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Richmond, Virginia

REFERENCES:
- [Derived] Strezova A, Lal H, Enweonye I, Campora L, Beukelaers P, Segall N, Heineman TC, Schuind AE, Oostvogels L. The adjuvanted recombinant zoster vaccine co-administered with a tetanus, diphtheria and pertussis vaccine in adults aged >/=50 years: A randomized trial. Vaccine. 2019 Sep 16;37(39):5877-5885. doi: 10.1016/j.vaccine.2019.08.001. Epub 2019 Aug 20. PMID 31443993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not all subjects who were enrolled started the study due to elimination from statistical analyses or no vaccination received.
Pre-assignment Details: For one subject, the reason for withdrawal was incorrectly entered into the eCRF as "lost due to Crohn's disease." The subject withdrew from the study due to a combination of irritable bowel syndrome and time constraints associated with employment. This information was clarified after database freeze.
Period: Active Phase
Arm/Group | GSK1437173A Group | Control Group
Started | 412 | 418
Completed | 396 | 398
Not Completed | 16 | 20
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 8 | 11
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Enrolled in error | 1 | 0
Not completed — Lost due to Crohn's disease | 0 | 1
Period: Safety Phase
Arm/Group | GSK1437173A Group | Control Group
Started | 412 | 418
Completed | 385 | 383
Not Completed | 27 | 35
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 11 | 18
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Enrolled in error | 1 | 0
Not completed — Lost due to Crohn's disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Control Group | Total
Number analyzed (Participants) | 412 | 418 | 830
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.4) | 63.1 (9.0) | 63.25 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 225 | 447
  Male | 190 | 193 | 383
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 41 | 53 | 94
  Geographic ancestry: American Indian or Alaskan Native | 1 | 1 | 2
  Geographic ancestry: Asian - Central/South Asian Heritage | 0 | 1 | 1
  Geographic ancestry: Asian - East Asian Heritage | 0 | 1 | 1
  Geographic ancestry: Asian - Japanese Heritage | 1 | 0 | 1
  Geographic ancestry: White - Arabic/North African Heritage | 3 | 0 | 3
  Geographic ancestry: White - Caucasian/European Heritage | 364 | 357 | 721
  Geographic ancestry: Mixed Origin | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Vaccine Response for Anti-glycoprotein E (Anti-gE) in GSK1437173A Group
Description: This outcome was required only for the GSK1437173A Group. Vaccine response defined as:
  For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL); For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: At 1 month post-Dose 2 (Month 3)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included subjects meeting all eligibility criteria for whom data concerning immunogenicity endpoint measures were available, only for subjects in the GSK1437173A Group.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 369
Participants | 361

2. Primary Outcome: Antibody Concentrations Against Glycoprotein E (Anti-gE)
Description: Antibody concentrations against glycoprotein E (gE) have been assessed by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The reference seropositivity cut-off was an anti-gE antibody concentration greater than or equal to (≥) 97 mIU/mL.
Time Frame: At 1 month post-Dose 2 (Month 3 for GSK1437173A Group adn Month 5 for Control Group)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included subjects meeting all eligibility criteria for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 369 | 380
mIU/mL | 51687.7 [48425.1 to 55170.1] | 57998.6 [54456.9 to 61770.6]
Statistical Analysis 1: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to two doses of the GSK1437173A vaccine when Boostrix vaccine was co-administered with the first GSK1437173A vaccine dose compared to two doses of GSK1437173A vaccine (administered separately from Boostrix vaccine), one month after the last vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the last vaccine dose (Month 3 or Month 5), the upper limit (UL) of the 95% confidence interval (CI) for the anti-gE antibodies GMC ratio between the Control Group and the GSK1437173A Group had to be below (<) 1.5,; Adjustment for baseline concentration and age - pooled variance; Adjusted GMC ratio = 1.11, 95% CI 2-sided [1.02 to 1.21]

3. Primary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN) Antigens
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations have been assessed by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: At 1 month post-Dose 1 (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 374 | 394
IU/mL
  Anti-PT | 41.1 [36.2 to 46.7] | 53.9 [47.4 to 61.4]
  Anti-FHA: number analyzed (Participants) | 373 | 391
  Anti-FHA | 309.3 [276.4 to 346.0] | 399.4 [359.1 to 444.3]
  Anti-PRN: number analyzed (Participants) | 370 | 392
  Anti-PRN | 222.6 [186.3 to 266.0] | 278.1 [232.9 to 332.0]
Statistical Analysis 1: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to Boostrix vaccine when co-administered with GSK1437173A vaccine at first vaccination dose compared to Boostrix vaccine (administered separately from GSK1437173A) for pertussis toxoid (PT), one month after the vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the first vaccine dose (Month 1), the upper limit (UL) of the 95% confidence interval for the GMC ratio for anti-PT antibodies of the Control Group over the GSK1437173A Group had to be < 1.5; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 1.17, 95% CI 2-sided [1.00 to 1.36]
Statistical Analysis 2: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to Boostrix vaccine when co-administered with GSK1437173A vaccine at first vaccination dose compared to Boostrix vaccine (administered separately from GSK1437173A) for filamentous hemagglutinin (FHA) antigen, one month after the vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the first vaccine dose (Month 1), the upper limit (UL) of the 95% confidence interval for the GMC ratio for anti-FHA antibodies of the Control Group over the GSK1437173A Group had to be < 1.5; Adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 1.24, 95% CI 2-sided [1.07 to 1.44]
Statistical Analysis 3: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to Boostrix vaccine when co-administered with GSK1437173A vaccine at first vaccination dose compared to Boostrix vaccine (administered separately from GSK1437173A) for pertactin (PRN) antigen, one month after the vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the first vaccine dose (Month 1), the upper limit (UL) of the 95% confidence interval for the GMC ratio for anti-PRN antibodies of the Control Group over the GSK1437173A Group had to be < 1.5; Adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 1.27, 95% CI 2-sided [1.02 to 1.58]

4. Primary Outcome: Antibody Concentrations Against Diphteria (Anti-D) and Tetanus (Anti-T) Antigens
Description: as for outcome 3
Time Frame: At 1 month post-Dose 1 (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 374 | 394
IU/mL
  Anti-D: number analyzed (Participants) | 374 | 389
  Anti-D | 2.2 [1.9 to 2.6] | 2.5 [2.1 to 3.0]
  Anti-T | 8.7 [7.8 to 9.7] | 10.1 [9.0 to 11.4]
Statistical Analysis 1: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to Boostrix vaccine when co-administered with GSK1437173A vaccine at first vaccination dose compared to Boostrix vaccine (administered separately from GSK1437173A) for diphteria (D) antigen, one month after the vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the first vaccine dose (Month 1), the upper limit (UL) of the 95% confidence interval (CI) for the difference in the percentages of subjects with anti-diphtheria (anti-D) concentrations ≥ 1.0 IU/mL of the Control Group minus the GSK1437173A Group had to be < 10%; Difference in seropositivity rate = -0.10, 95% CI 2-sided [-3.03 to 2.85]
Statistical Analysis 2: Comparison: GSK1437173A Group vs Control Group; Demonstration of non-inferiority of the humoral immune response to Boostrix vaccine when co-administered with GSK1437173A vaccine at first vaccination dose compared to Boostrix vaccine (administered separately from GSK1437173A) for tetanus (T) antigen, one month after the vaccine dose; Test type: Non-Inferiority — Criteria for non-inferiority: At one month after the first vaccine dose (Month 1), the upper limit (UL) of the 95% confidence interval (CI) for the difference in the percentages of subjects with anti-tetanus (anti-T) concentrations ≥ 1.0 IU/mL of the Control Group minus the GSK1437173A Group had to be < 10%; Difference in seropositivity rate = 0.01, 95% CI 2-sided [-1.18 to 1.27]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, by Dose
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond (>) 100 millimeters (mm).
  "0" Implied that no data was applicable for the GSK1437173A Group at Dose 3, since it received only 2 vaccine doses
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented, on subjects with their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 407 | 412
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 407 | 409
  Any Pain, Dose 1 | 315 | 156
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Pain, Dose 1 | 26 | 3
  Any Redness, Dose 1: number analyzed (Participants) | 407 | 409
  Any Redness, Dose 1 | 119 | 18
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Redness, Dose 1 | 1 | 1
  Any Swelling, Dose 1: number analyzed (Participants) | 407 | 409
  Any Swelling, Dose 1 | 79 | 22
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Swelling, Dose 1 | 1 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 390 | 403
  Any Pain, Dose 2 | 289 | 299
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Pain, Dose 2 | 15 | 21
  Any Redness, Dose 2: number analyzed (Participants) | 390 | 403
  Any Redness, Dose 2 | 116 | 102
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Redness, Dose 2 | 5 | 3
  Any Swelling, Dose 2: number analyzed (Participants) | 390 | 403
  Any Swelling, Dose 2 | 83 | 67
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Swelling, Dose 2 | 1 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 395
  Any Pain, Dose 3 | 0 | 282
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Pain, Dose 3 | 0 | 24
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 395
  Any Redness, Dose 3 | 0 | 101
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Redness, Dose 3 | 0 | 3
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 395
  Any Swelling, Dose 3 | 0 | 76
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across doses | 346 | 357
  Grade 3 Pain, Across doses | 39 | 39
  Any Redness, Across doses | 167 | 148
  Grade 3 Redness, Across doses | 6 | 7
  Any Swelling, Across doses | 124 | 115
  Grade 3 Swelling, Across doses | 2 | 1

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, by Study Vaccine
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond (>) 100 millimeters (mm).
  "0" implies that: 1. No data were applicable for the GSK1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group 2. No data were applicable for the Boostrix vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for both the groups.
  3. No data were applicable for the GSK1437173A Group at Dose 3, since it received only 2 vaccine doses.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 407 | 409
Participants
  Any Pain, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Any Pain, Boostrix vaccine, Dose 1 | 183 | 156
  Grade 3 Pain, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Grade 3 Pain, Boostrix vaccine, Dose 1 | 8 | 3
  Any Pain, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Any Pain, GSK1437173A vaccine, Dose 1 | 290 | 0
  Grade 3 Pain, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Grade 3 Pain, GSK1437173A vaccine, Dose 1 | 20 | 0
  Any Redness, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Any Redness, Boostrix vaccine, Dose 1 | 31 | 18
  Grade 3 Redness, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Grade 3 Redness, Boostrix vaccine, Dose 1 | 0 | 1
  Any Redness, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Any Redness, GSK1437173A vaccine, Dose 1 | 108 | 0
  Grade 3 Redness, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Grade 3 Redness, GSK1437173A vaccine, Dose 1 | 1 | 0
  Any Swelling, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Any Swelling, Boostrix vaccine, Dose 1 | 23 | 22
  Grade 3 Swelling, Boostrix vaccine, Dose 1: number analyzed (Participants) | 406 | 409
  Grade 3 Swelling, Boostrix vaccine, Dose 1 | 0 | 1
  Any Swelling, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Any Swelling, GSK1437173A vaccine, Dose 1 | 67 | 0
  Grade 3 Swelling, GSK1437173A vaccine, Dose 1: number analyzed (Participants) | 407 | 0
  Grade 3 Swelling, GSK1437173A vaccine, Dose 1 | 1 | 0
  Any Pain, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Any Pain, Boostrix vaccine, Dose 2 | 0 | 0
  Grade 3 Pain, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Grade 3 Pain, Boostrix vaccine, Dose 2 | 0 | 0
  Any Pain, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Any Pain, GSK1437173A vaccine, Dose 2 | 289 | 299
  Grade 3 Pain, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Pain, GSK1437173A vaccine, Dose 2 | 15 | 21
  Any Redness, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Any Redness, Boostrix vaccine, Dose 2 | 0 | 0
  Grade 3 Redness, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Grade 3 Redness, Boostrix vaccine, Dose 2 | 0 | 0
  Any Redness, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Any Redness, GSK1437173A vaccine, Dose 2 | 116 | 102
  Grade 3 Redness, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Redness, GSK1437173A vaccine, Dose 2 | 5 | 3
  Any Swelling, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Any Swelling, Boostrix vaccine, Dose 2 | 0 | 0
  Grade 3 Swelling, Boostrix vaccine, Dose 2: number analyzed (Participants) | 0 | 0
  Grade 3 Swelling, Boostrix vaccine, Dose 2 | 0 | 0
  Any Swelling, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Any Swelling, GSK1437173A vaccine, Dose 2 | 83 | 67
  Grade 3 Swelling, GSK1437173A vaccine, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Swelling, GSK1437173A vaccine, Dose 2 | 1 | 0
  Any Pain, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Any Pain, Boostrix vaccine, Dose 3 | 0 | 0
  Grade 3 Pain, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Grade 3 Pain, Boostrix vaccine, Dose 3 | 0 | 0
  Any Pain, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Any Pain, GSK1437173A vaccine, Dose 3 | 0 | 282
  Grade 3 Pain, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Pain, GSK1437173A vaccine, Dose 3 | 0 | 24
  Any Redness, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Any Redness, Boostrix vaccine, Dose 3 | 0 | 0
  Grade 3 Redness, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Grade 3 Redness, Boostrix vaccine, Dose 3 | 0 | 0
  Any Redness, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Any Redness, GSK1437173A vaccine, Dose 3 | 0 | 101
  Grade 3 Redness, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Redness, GSK1437173A vaccine, Dose 3 | 0 | 3
  Any Swelling, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Any Swelling, Boostrix vaccine, Dose 3 | 0 | 0
  Grade 3 Swelling, Boostrix vaccine, Dose 3: number analyzed (Participants) | 0 | 0
  Grade 3 Swelling, Boostrix vaccine, Dose 3 | 0 | 0
  Any Swelling, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Any Swelling, GSK1437173A vaccine, Dose 3 | 0 | 76
  Grade 3 Swelling, GSK1437173A vaccine, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Swelling, GSK1437173A vaccine, Dose 3 | 0 | 0
  Any Pain, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Any Pain, Boostrix vaccine, Across doses | 183 | 156
  Grade 3 Pain, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Grade 3 Pain, Boostrix vaccine, Across doses | 8 | 3
  Any Pain, GSK1437173A vaccine, Across doses: number analyzed (Participants) | 407 | 403
  Any Pain, GSK1437173A vaccine, Across doses | 339 | 344
  Grade 3 Pain, GSK1437173A vaccine, Across doses: number analyzed (Participants) | 407 | 403
  Grade 3 Pain, GSK1437173A vaccine, Across doses | 34 | 37
  Any Redness, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Any Redness, Boostrix vaccine, Across doses | 31 | 18
  Grade 3 Redness, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Grade 3 Redness, Boostrix vaccine, Across doses | 0 | 1
  Any Redness, GSK1437173A vaccine, Across doses: number analyzed (Participants) | 407 | 403
  Any Redness, GSK1437173A vaccine, Across doses | 163 | 144
  Grade 3 Redness, GSK1437173A vaccine, Across doses: number analyzed (Participants) | 407 | 403
  Grade 3 Redness, GSK1437173A vaccine, Across doses | 6 | 6
  Any Swelling, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Any Swelling, Boostrix vaccine, Across doses | 23 | 22
  Grade 3 Swelling, Boostrix vaccine, Across doses: number analyzed (Participants) | 406 | 409
  Grade 3 Swelling, Boostrix vaccine, Across doses | 0 | 1
  Any Swelling, GSK1437173A vaccine, Across doses: number analyzed (Participants) | 407 | 403
  Any Swelling, GSK1437173A vaccine, Across doses | 117 | 109
  Grade 3 Swelling, GSK1437173A vaccine,Across doses: number analyzed (Participants) | 407 | 403
  Grade 3 Swelling, GSK1437173A vaccine,Across doses | 2 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms, by Dose
Description: Assessed solicited general symptoms were fatigue, gastrointestinal (symptoms included nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia, shivering and fever [defined as oral, axillary, rectal or tympanic temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = temperature above (>) 39.0 °C. Related = general symptom assessed by the investigator as causally related to vaccination.
  "0" Implied that no data was applicable for the GSK1437173A Group at Dose 3, since it received only 2 vaccine doses
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analisys was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented, on subjects with their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 407 | 412
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 407 | 409
  Any Fatigue, Dose 1 | 129 | 65
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Fatigue, Dose 1 | 12 | 7
  Related Fatigue, Dose 1: number analyzed (Participants) | 407 | 409
  Related Fatigue, Dose 1 | 88 | 37
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 407 | 409
  Any Gastrointestinal, Dose 1 | 52 | 35
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Gastrointestinal, Dose 1 | 2 | 3
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 407 | 409
  Related Gastrointestinal, Dose 1 | 25 | 16
  Any Headache, Dose 1: number analyzed (Participants) | 407 | 409
  Any Headache, Dose 1 | 106 | 60
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Headache, Dose 1 | 7 | 3
  Related Headache, Dose 1: number analyzed (Participants) | 407 | 409
  Related Headache, Dose 1 | 74 | 32
  Any Myalgia, Dose 1: number analyzed (Participants) | 407 | 409
  Any Myalgia, Dose 1 | 177 | 102
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Myalgia, Dose 1 | 12 | 4
  Related Myalgia, Dose 1: number analyzed (Participants) | 407 | 409
  Related Myalgia, Dose 1 | 134 | 76
  Any Shivering, Dose 1: number analyzed (Participants) | 407 | 409
  Any Shivering, Dose 1 | 64 | 16
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Shivering, Dose 1 | 6 | 3
  Related Shivering, Dose 1: number analyzed (Participants) | 407 | 409
  Related Shivering, Dose 1 | 48 | 8
  Any Temperature, Dose 1: number analyzed (Participants) | 407 | 409
  Any Temperature, Dose 1 | 36 | 7
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 407 | 409
  Grade 3 Temperature, Dose 1 | 2 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 407 | 409
  Related Temperature, Dose 1 | 26 | 5
  Any Fatigue, Dose 2: number analyzed (Participants) | 390 | 403
  Any Fatigue, Dose 2 | 137 | 110
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Fatigue, Dose 2 | 22 | 9
  Related Fatigue, Dose 2: number analyzed (Participants) | 390 | 403
  Related Fatigue, Dose 2 | 101 | 74
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 390 | 403
  Any Gastrointestinal, Dose 2 | 51 | 46
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Gastrointestinal, Dose 2 | 5 | 5
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 390 | 403
  Related Gastrointestinal, Dose 2 | 34 | 28
  Any Headache, Dose 2: number analyzed (Participants) | 390 | 403
  Any Headache, Dose 2 | 99 | 82
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Headache, Dose 2 | 10 | 8
  Related Headache, Dose 2: number analyzed (Participants) | 390 | 403
  Related Headache, Dose 2 | 74 | 54
  Any Myalgia, Dose 2: number analyzed (Participants) | 390 | 403
  Any Myalgia, Dose 2 | 160 | 155
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Myalgia, Dose 2 | 17 | 16
  Related Myalgia, Dose 2: number analyzed (Participants) | 390 | 403
  Related Myalgia, Dose 2 | 122 | 116
  Any Shivering, Dose 2: number analyzed (Participants) | 390 | 403
  Any Shivering, Dose 2 | 79 | 38
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Shivering, Dose 2 | 12 | 4
  Related Shivering, Dose 2: number analyzed (Participants) | 390 | 403
  Related Shivering, Dose 2 | 60 | 27
  Any Temperature, Dose 2: number analyzed (Participants) | 390 | 403
  Any Temperature, Dose 2 | 51 | 23
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 390 | 403
  Grade 3 Temperature, Dose 2 | 2 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 390 | 403
  Related Temperature, Dose 2 | 32 | 16
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 395
  Any Fatigue, Dose 3 | 0 | 130
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Fatigue, Dose 3 | 0 | 14
  Related Fatigue, Dose 3: number analyzed (Participants) | 0 | 395
  Related Fatigue, Dose 3 | 0 | 92
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 0 | 395
  Any Gastrointestinal, Dose 3 | 0 | 54
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Gastrointestinal, Dose 3 | 0 | 3
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 0 | 395
  Related Gastrointestinal, Dose 3 | 0 | 37
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 395
  Any Headache, Dose 3 | 0 | 95
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Headache, Dose 3 | 0 | 8
  Related Headache, Dose 3: number analyzed (Participants) | 0 | 395
  Related Headache, Dose 3 | 0 | 69
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 395
  Any Myalgia, Dose 3 | 0 | 164
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Myalgia, Dose 3 | 0 | 19
  Related Myalgia, Dose 3: number analyzed (Participants) | 0 | 395
  Related Myalgia, Dose 3 | 0 | 124
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 395
  Any Shivering, Dose 3 | 0 | 65
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Shivering, Dose 3 | 0 | 11
  Related Shivering, Dose 3: number analyzed (Participants) | 0 | 395
  Related Shivering, Dose 3 | 0 | 50
  Any Temperature, Dose 3: number analyzed (Participants) | 0 | 395
  Any Temperature, Dose 3 | 0 | 43
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 0 | 395
  Grade 3 Temperature, Dose 3 | 0 | 1
  Related Temperature, Dose 3: number analyzed (Participants) | 0 | 395
  Related Temperature, Dose 3 | 0 | 28
  Any Fatigue, Across doses | 186 | 192
  Grade 3 Fatigue, Across doses | 30 | 27
  Related Fatigue, Across doses | 143 | 134
  Any Gastrointestinal, Across doses | 85 | 97
  Grade 3 Gastrointestinal, Across doses | 7 | 9
  Related Gastrointestinal, Across doses | 51 | 62
  Any Headache, Across doses | 152 | 158
  Grade 3 Headache, Across doses | 16 | 15
  Related Headache, Across doses | 118 | 108
  Any Myalgia, Across doses | 227 | 243
  Grade 3 Myalgia, Across doses | 27 | 32
  Related Myalgia, Across doses | 176 | 186
  Any Shivering, Across doses | 112 | 100
  Grade 3 Shivering, Across doses | 18 | 16
  Related Shivering, Across doses | 86 | 72
  Any Temperature, Across doses | 72 | 63
  Grade 3 Temperature, Across doses | 3 | 1
  Related Temperature, Across doses | 48 | 41

8. Secondary Outcome: Number of Days With Solicited Symptoms
Description: The number of days with local and general symptoms have been assessed during the solicited post-vaccination period.
  "0" Implied that no data was applicable for the GSK1437173A Group at Dose 3, since it received only 2 vaccine doses
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 7
Measure: Mean (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 407 | 409
Number analyzed (Doses with the symptom) | 315 | 299
Days
  Pain, Dose 1: number analyzed (Doses with the symptom) | 315 | 156
  Pain, Dose 1 | 3.2 [2.0 to 4.0] | 2.6 [2.0 to 3.0]
  Pain, Dose 2: number analyzed (Participants) | 390 | 403
  Pain, Dose 2: number analyzed (Doses with the symptom) | 289 | 299
  Pain, Dose 2 | 2.8 [2.0 to 4.0] | 2.9 [2.0 to 4.0]
  Pain, Dose 3: number analyzed (Participants) | 0 | 395
  Pain, Dose 3: number analyzed (Doses with the symptom) | 0 | 282
  Pain, Dose 3 |  | 2.7 [2.0 to 3.0]
  Redness, Dose 1: number analyzed (Doses with the symptom) | 119 | 18
  Redness, Dose 1 | 3.3 [2.0 to 5.0] | 3.0 [2.0 to 5.0]
  Redness, Dose 2: number analyzed (Participants) | 390 | 403
  Redness, Dose 2: number analyzed (Doses with the symptom) | 116 | 102
  Redness, Dose 2 | 3.2 [2.0 to 4.0] | 3.2 [2.0 to 4.0]
  Redness, Dose 3: number analyzed (Participants) | 0 | 395
  Redness, Dose 3: number analyzed (Doses with the symptom) | 0 | 101
  Redness, Dose 3 |  | 2.9 [2.0 to 4.0]
  Swelling, Dose 1: number analyzed (Doses with the symptom) | 79 | 22
  Swelling, Dose 1 | 3.3 [2.0 to 5.0] | 3.5 [2.0 to 5.0]
  Swelling, Dose 2: number analyzed (Participants) | 390 | 403
  Swelling, Dose 2: number analyzed (Doses with the symptom) | 83 | 67
  Swelling, Dose 2 | 3.1 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Swelling, Dose 3: number analyzed (Participants) | 0 | 395
  Swelling, Dose 3: number analyzed (Doses with the symptom) | 0 | 76
  Swelling, Dose 3 |  | 2.9 [2.0 to 4.0]
  Fatigue, Dose 1: number analyzed (Doses with the symptom) | 129 | 65
  Fatigue, Dose 1 | 2.4 [1.0 to 3.0] | 2.5 [1.0 to 4.0]
  Fatigue, Dose 2: number analyzed (Participants) | 390 | 403
  Fatigue, Dose 2: number analyzed (Doses with the symptom) | 137 | 110
  Fatigue, Dose 2 | 2.3 [1.0 to 3.0] | 2.7 [1.0 to 3.0]
  Fatigue, Dose 3: number analyzed (Participants) | 0 | 395
  Fatigue, Dose 3: number analyzed (Doses with the symptom) | 0 | 130
  Fatigue, Dose 3 |  | 2.6 [1.0 to 4.0]
  Gastrointestinal, Dose 1: number analyzed (Doses with the symptom) | 52 | 35
  Gastrointestinal, Dose 1 | 2.3 [1.0 to 4.0] | 2.1 [1.0 to 3.0]
  Gastrointestinal, Dose 2: number analyzed (Participants) | 390 | 403
  Gastrointestinal, Dose 2: number analyzed (Doses with the symptom) | 51 | 46
  Gastrointestinal, Dose 2 | 2.0 [1.0 to 2.0] | 2.3 [1.0 to 3.0]
  Gastrointestinal, Dose 3: number analyzed (Participants) | 0 | 395
  Gastrointestinal, Dose 3: number analyzed (Doses with the symptom) | 0 | 54
  Gastrointestinal, Dose 3 |  | 1.9 [1.0 to 3.0]
  Headache, Dose 1: number analyzed (Doses with the symptom) | 106 | 60
  Headache, Dose 1 | 1.8 [1.0 to 2.0] | 2.2 [1.0 to 2.0]
  Headache, Dose 2: number analyzed (Participants) | 390 | 403
  Headache, Dose 2: number analyzed (Doses with the symptom) | 99 | 82
  Headache, Dose 2 | 1.9 [1.0 to 2.0] | 2.1 [1.0 to 3.0]
  Headache, Dose 3: number analyzed (Participants) | 0 | 395
  Headache, Dose 3: number analyzed (Doses with the symptom) | 0 | 95
  Headache, Dose 3 |  | 2.0 [1.0 to 2.0]
  Myalgia, Dose 1: number analyzed (Doses with the symptom) | 177 | 102
  Myalgia, Dose 1 | 2.9 [2.0 to 4.0] | 2.3 [1.0 to 3.0]
  Myalgia, Dose 2: number analyzed (Participants) | 390 | 403
  Myalgia, Dose 2: number analyzed (Doses with the symptom) | 160 | 155
  Myalgia, Dose 2 | 2.7 [2.0 to 3.5] | 2.9 [1.0 to 4.0]
  Myalgia, Dose 3: number analyzed (Participants) | 0 | 395
  Myalgia, Dose 3: number analyzed (Doses with the symptom) | 0 | 164
  Myalgia, Dose 3 |  | 2.7 [1.0 to 3.0]
  Shivering, Dose 1: number analyzed (Doses with the symptom) | 64 | 16
  Shivering, Dose 1 | 1.6 [1.0 to 2.0] | 2.3 [1.0 to 3.0]
  Shivering, Dose 2: number analyzed (Participants) | 390 | 403
  Shivering, Dose 2: number analyzed (Doses with the symptom) | 79 | 38
  Shivering, Dose 2 | 1.6 [1.0 to 2.0] | 1.6 [1.0 to 2.0]
  Shivering, Dose 3: number analyzed (Participants) | 0 | 395
  Shivering, Dose 3: number analyzed (Doses with the symptom) | 0 | 65
  Shivering, Dose 3 |  | 1.5 [1.0 to 1.0]
  Temperature, Dose 1: number analyzed (Doses with the symptom) | 36 | 7
  Temperature, Dose 1 | 1.7 [1.0 to 2.0] | 2.4 [1.0 to 3.0]
  Temperature, Dose 2: number analyzed (Participants) | 390 | 403
  Temperature, Dose 2: number analyzed (Doses with the symptom) | 51 | 23
  Temperature, Dose 2 | 1.6 [1.0 to 2.0] | 1.5 [1.0 to 1.0]
  Temperature, Dose 3: number analyzed (Participants) | 0 | 395
  Temperature, Dose 3: number analyzed (Doses with the symptom) | 0 | 43
  Temperature, Dose 3 |  | 1.5 [1.0 to 2.0]

9. Secondary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related = pIMDs assessed by the investigator as causally related to the study vaccination.
Time Frame: From first vaccination up to study end (Day 0 to Month 14)
Population: The analisys was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 412 | 418
Participants
  Any pIMD(s) | 0 | 0
  Related pIMD(s) | 0 | 0

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 412 | 418
Participants
  Any AE(s) | 105 | 118
  Grade 3 AE(s) | 10 | 15
  Related AE(s) | 27 | 31

11. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination up to study end (Day 0 to Month 14)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 412 | 418
Participants | 21 | 31

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 30-day (Days 0-29) post-vaccination period; SAEs: from first vaccination up to study end at Month 14.
Arm/Group | GSK1437173A Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/412 | 5/418
Serious Adverse Events (participants affected / at risk) | 21/412 | 31/418
Other Adverse Events (participants affected / at risk) | 368/412 | 380/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=412) | Control Group (N=418)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Surgical failure (General disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Device failure (Product Issues) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=412) | Control Group (N=418)
Chills (General disorders) | 112 (144) | 102 (121)
Erythema (Skin and subcutaneous tissue disorders) | 167 (235) | 148 (222)
Fatigue (General disorders) | 186 (267) | 192 (306)
Gastrointestinal disorder (Gastrointestinal disorders) | 85 (103) | 97 (135)
Headache (Nervous system disorders) | 153 (207) | 159 (242)
Myalgia (Musculoskeletal and connective tissue disorders) | 228 (341) | 243 (423)
Pain (General disorders) | 346 (605) | 357 (740)
Pyrexia (General disorders) | 74 (89) | 64 (76)
Swelling (General disorders) | 124 (162) | 115 (165)

LIMITATIONS AND CAVEATS:
At the time of posting this record, only the safety and demography results until 1-month post-last vaccination (Co-ad group Month 3 and Control group Month 5) were available. The record will be updated once immunogenicity results become available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.